CLINICAL TRIAL: NCT03123068
Title: Cocoa Flavanols for Modulating the Surgical Immune Response and Accelerating Clinical Recovery
Brief Title: Cocoa Flavanols for Modulating Immune Response and Accelerating Recovery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Martin Angst, Professor of Anethesioloogy, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 39535
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Surgical Recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo and active treatments will be formulated in identical capsules, and bottled and labeled with coded study numbers that will allow for all parties to remain blinded throughout the data collection phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active treatment group - Group A (Active Comparator): Participants will receive a daily oral dose of 1,000 mg cocoa flavanol (CocoaVia®) for 5 days before surgery. The daily dose will consist of 8 capsules in divided doses throughout the day.
  Interventions: Drug: CocoaVia®
- Placebo treatment group - Group B (Placebo Comparator): Participants will receive a daily oral dose of a placebo for 5 days before surgery. The daily dose will consist of 8 capsules in divided doses throughout the day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CocoaVia® — CocoaVia® is manufactured by Mars, Inc. It is a dietary supplement of cocoa bean extract, containing 125 mg cocoa flavanols per capsule.
  Other Names: Cocoa flavanol
  Arms: Active treatment group - Group A
Other: Placebo — The placebo capsules will contain an inert ingredient packaged to be indistinguishable from the active treatment.
  Arms: Placebo treatment group - Group B

SUMMARY:
This double-blind, placebo-controlled proof-of-concept clinical trial is intended to demonstrate that preemptive oral administration of cocoa flavanol for five days before surgery will attenuate the surgery-evoked increase of HMGB1 in blood plasma and NFkB signaling in innate immune cells shortly after surgery. A secondary aim is to capture preliminary patient-centered outcomes data and relate these outcomes to the intake of oral cocoa flavanol and surgery-evoked activation of the HMGB1-NFkB signaling axis. Participants will be randomized to receive either an over the counter supplement containing cocoa flavanols, or placebo, for 5 days before surgery.

DETAILED DESCRIPTION:
During the last two decades significant effort has been made to enhance recovery after surgery. Despite the implementation of pragmatic and standardized clinical protocols to enhance recovery and shorten hospital length of stay, the utility of these protocols for improving patient-centered recovery cost-effectively remains uncertain. Critical elements of recovery that greatly matter to patients and health care providers include the resolution of pain, daily functioning, and loss of postoperative fatigue. A patient-centered and cost-effective focus on postoperative recovery pays tribute to three goals of health care: Improving patients' experience, improving health, and constraining per capita cost. As such, novel and cost-effective strategies are greatly needed to accelerate patient-recovery after surgery.

Preliminary data by Dr. Angst and his collaborators indicate that administration of a cocoa flavanol extract that is equivalent in dose to the amount of cocoa flavanol contained in about 50 grams of dark chocolate decreases plasma levels of HMGB1. HMGB1 is an archetypical alarmin, i.e., an endogenous mediator that is released upon cellular stress and injury. HMGB1 triggers a pro-inflammatory cascade by binding to toll-like receptors (TLRs) on innate immune and other cells, which results in activation of pro-inflammatory transcription factors (e.g. NFkB) and the subsequent release of major pro-inflammatory cytokines (e.g. TNFα). The prominent role of the HMGB1-TLR axis in inflammatory disease states including surgery, trauma, stroke, and myocardial infarction has recently been highlighted.16-19 Importantly, dampening activity along this pathway in preclinical injury models has been shown to improve outcomes.

The potential of HMGB1 as a therapeutic target in acute inflammatory disease states has recently been emphasized. A major challenge is the identification of effective and non-toxic clinical strategies that can safely modulate HMGB1 in humans. This research study will evaluate a safe, highly scalable, and relatively cheap pre-surgical nutritional intervention that has significant potential to do just that, safely modulate HMGB1 and improve clinical recovery after surgery. As such, this proposed research could change clinical practice within years. While studied intervention targets a specific pro-inflammatory pathway implicated in aggravated tissue damage and delayed healing/recovery, the use of broader and less specific anti-inflammatory interventions in the perioperative period including non-steroidal anti-inflammatory drugs and corticosteroids is common clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 90 years of age
2. Male or female
3. Planning to undergo total hip or knee arthroplasty, either primary or revision
4. Fluent in English
5. Willing and able to sign an informed consent form and HIPAA authorization and to comply with study procedures

Exclusion Criteria:

1. Infectious disease within the last month
2. Immune-suppressant therapy within the last 2 months (e.g., azathioprine or cyclosporine)
3. Chronic medication with potential immune-modulatory effects (e.g., daily oral morphine-equivalent intake > 30 mg)
4. Major surgery within the last 3 months or minor surgery within the last month.
5. History of substance abuse (e.g., alcoholism, drug dependency)
6. Pregnancy
7. Autoimmune disease interfering with data interpretation (e.g. lupus)
8. Renal, hepatic, cardiovascular, or respiratory diseases resulting in clinically relevant impaired function
9. Active malignancy
10. Participation in another clinical trial of an investigational drug or device within the last month that, in the investigator's opinion, would create an increased risk to the participant or compromise the integrity of the study
11. Other conditions compromising a participant's safety or the integrity of the study
12. Allergy to active ingredient of CocoaVia®, the study intervention.
13. Frequent consumption of dark chocolate and flavanol containing foods (e.g. black tea, red wine, apples)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in the pre-anesthesia and orthopedic clinics at Stanford Medical Center. Recruitment was conducted from 3/01/2017 with the final study intervention for the final patient on 12/14/2018.
Pre-assignment Details: A total of 32 participants that were consented/enrolled were dropped prior to randomization for a variety of reasons. Participants changed their minds, exclusion criteria were identified after consent but before study participation began, and early non-compliance with the survey completion were all reasons for withdrawal after consent.
Period: Overall Study
Arm/Group | Active Treatment Group - Group A | Placebo Treatment Group - Group B
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment Group - Group A | Placebo Treatment Group - Group B | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 20
  >=65 years | 14 | 8 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 18 | 16 | 34
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 13 | 32
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: NFkB Signaling in Innate Immune Cells
Description: Blood samples will be collected to measure possible attenuation of surgery-evoked increase in NFkB signaling in innate immune cells shortly after surgery at specified time points.
  Phosphorylation of functional markers (activity) was expressed as the arcsinh-transformed value of the median value. Changes in activity over time were captured by building the arcsinh ratio between the arcsinh-value obtained in samples collected at a given time with the arcsinh-value obtained in samples collected at baseline, i.e., before starting the intervention with CocoaVia. Results are reported for NFkB (p65).
Time Frame: 1 hour and 48 hours following surgery
Population: Participants with available data are included in the analysis.
  Three patients were excluded from the molecular analysis because of incorrect intake of the study medication, difficulties obtaining blood draws, and a non-recognized immune disorder. Exclusion of patients from the analyses was determined before unblinding.
Measure: Median (Inter-Quartile Range); unit: NFkB (p65) arcsinh ratio
Arm/Group | Active Treatment Group - Group A | Placebo Treatment Group - Group B
Number analyzed (Participants) | 20 | 19
NFkB (p65) arcsinh ratio
  1 hour following surgery | 0.68 [0.41 to 0.80] | 0.69 [0.53 to 0.79]
  48 hours following surgery | 0.71 [0.44 to 0.81] | 0.71 [0.59 to 0.85]

2. Secondary Outcome: HMGB1 Level in Blood Plasma
Description: Blood samples will be collected to measure possible attenuation of surgery-evoked increase of HMGB1 in blood plasma shortly after surgery at specified time points.
Time Frame: 1 hour and 48 hours following surgery.
Population: Three patients were excluded from the molecular analysis because of incorrect intake of the study medication, difficulties obtaining blood draws, and a non-recognized immune disorder. Four additional patients were excluded from the analysis including clinical data because respective questionnaires were not answered reliably. The total participants included in this analysis is 35. Exclusion of patients from the analyses was determined before unblinding.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Active Treatment Group - Group A | Placebo Treatment Group - Group B
Number analyzed (Participants) | 17 | 18
ng/ml
  1 hour following surgery | NA [NA to NA] — Value below level of sensitivity for this assay. | NA [NA to NA] — Value below level of sensitivity for this assay.
  48 hours following surgery | NA [NA to NA] — Value below level of sensitivity for this assay. | NA [NA to NA] — Value below level of sensitivity for this assay.

3. Secondary Outcome: Step Count Per Minute as a Measure of Functional Recovery - Objective
Description: Participants wear an Actigraph watch with measurements taken every 30 seconds. The watch objectively and continuously reports a participant's activity and sleep.
Time Frame: post-surgical observation period (6 weeks)
Population: Participants with available data are included in the analysis.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Active Treatment Group - Group A | Placebo Treatment Group - Group B
Number analyzed (Participants) | 18 | 18
steps | 0.02 (0.05) | 0.04 (0.06)
Statistical Analysis 1: Comparison: Active Treatment Group - Group A vs Placebo Treatment Group - Group B; Test type: Other; p > 0.05, Mann Whitney U test

4. Secondary Outcome: Days to Mild Impairment as a Measure of Functional Recovery - Subjective
Description: Participants will complete the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire (function subscale) before surgery, daily during hospitalization, and weekly through week 6 post op.
  Higher WOMAC scores equate to greater functional limitations. Range of possible scores is 0 - 68
Time Frame: 5 days before surgery though 6 weeks post op.
Population: Three patients were excluded from the molecular analysis because of incorrect intake of the study medication, difficulties obtaining blood draws, and a non-recognized immune disorder. Four additional patients were excluded from the analysis including clinical data because respective questionnaires were not answered reliably. Exclusion of patients from the analyses was determined before unblinding.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Active Treatment Group - Group A | Placebo Treatment Group - Group B
Number analyzed (Participants) | 17 | 18
days | 35 [14 to 42] | 14 [7 to 35]

5. Secondary Outcome: Days to Mild Pain as Assessed by WOMAC Pain Scores
Description: Participants will complete the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire (pain subscale) before surgery, daily during hospitalization, and weekly through week 6 post op.
  Higher WOMAC scores equate to greater pain. Range of possible scores is 0 - 20.
Time Frame: 5 days before surgery though 6 weeks post op.
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Active Treatment Group - Group A | Placebo Treatment Group - Group B
Number analyzed (Participants) | 17 | 18
days | 28 [14 to 37] | 25 [3 to 28]

6. Secondary Outcome: Days to Half Max Recovery From Fatigue
Description: Participants will complete the Surgery Recovery Scale (SRS) questionnaire before surgery, daily during hospitalization, and weekly through week 6 post op to evaluate post op fatigue.
  Higher SRS scores reflect less fatigue, lower scores reflect greater fatigue. Total SRS score range from 17.81 to 100.
Time Frame: 5 days before surgery though 6 weeks post op.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Active Treatment Group - Group A | Placebo Treatment Group - Group B
Number analyzed (Participants) | 17 | 18
days | 14 [7 to 21] | 7 [3 to 14]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Active Treatment Group - Group A | Placebo Treatment Group - Group B
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/20
Other Adverse Events (participants affected / at risk) | 8/22 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment Group - Group A (N=22) | Placebo Treatment Group - Group B (N=20)
Pain (General disorders) | 1 (1) | 0 — Poorly controlled post op pain resulting in tachycardia and prolonged hospital stay.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment Group - Group A (N=22) | Placebo Treatment Group - Group B (N=20)
bladder pain (Renal and urinary disorders) | 0 | 1
blisters at wound site (Skin and subcutaneous tissue disorders) | 1 | 2
bursitis (Infections and infestations) | 0 | 2
dizziness (Nervous system disorders) | 0 | 1
elevated BP (Vascular disorders) | 0 | 1
labile BP (Vascular disorders) | 0 | 1
loss of appitite (Metabolism and nutrition disorders) | 2 | 0
lower extremity swelling (Vascular disorders) | 5 | 1
nausea (Gastrointestinal disorders) | 2 | 1
pain (General disorders) | 0 | 2
tachycardia (Cardiac disorders) | 1 | 1
urinary frequency (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT03123068/Prot_SAP_000.pdf